CLINICAL TRIAL: NCT03161951
Title: Differential Diagnostics of Etiology of Acute Infections Based on the Analysis of Expression of Activation Markers on the Surface of Peripheral Blood Monocytes and Neutrophils.
Brief Title: Differential Diagnostics of Etiology of Acute Infections
Status: Completed | Type: Observational
Sponsor: The Republican Research and Practical Center for Epidemiology and Microbiology (Other)
Responsible Party: Principal Investigator, Andrei Y. Hancharou, Head of the Laboratory for Immunology and Cellular Biotechnology,, The Republican Research and Practical Center for Epidemiology and Microbiology
Other Study IDs: RRPCEM_NMAT
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Intestinal Infectious Diseases; Neuroinfections
Keywords: acute Infections, flow cytometry, cell activation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neuroinfections: Patients with acute neuroinfections of bacterial and viral ethology.
- Intestinal Infectious Diseases: Patients with acute intestinal infectious diseases of bacterial and viral ethology.
- Control group: Control group of healthy persons

SUMMARY:
Method for diagnostics of the origin of infections (bacterial vs viral) based on the identification of activation markers of blood neutrophils and monocytes will be developed.

DETAILED DESCRIPTION:
During the study, method for diagnostics of the origin of infections (bacterial vs viral) based on the identification of activation markers of blood neutrophils and monocytes will be developed.This method will allow to make a diagnosis within an hour after blood sampling.

The expression of the following markers of activation will be studied using flow cytometry: CD11b, CD11c, CD13, CD16, CD32, CD35, CD38, CD62L, CD64, CD66b, CD88, CD284, HLA-ABC and HLA-DR.

ELIGIBILITY:
Inclusion Criteria:

* neuroinfections or acute intestinal infections;
* the possibility of blood sampling within a period of up to 24 hours from the moment of admission to hospital;
* less than 72 hours passed after the onset of the disease and until blood was collected;

Exclusion Criteria:

* refuse of patient to participate in the trial;
* more than 24 hours passed after the patient entered the hospital;
* the disease began more than 72 hours ago;
* concomitant severe acute and chronic diseases;
* malignant neoplasms, treatment at a time of less than 1 year, autoimmune diseases in the phase of exacerbation;
* pregnancy/lactation;
* HIV, Hepatites B/C;
* active tuberculosis;
* alcohol use disorder/drug addiction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the infectious departments of city hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the diagnosis of bacterial vs viral acute infection | 1 month
  Sensitivity of the diagnosis of bacterial vs viral acute infection using proposed method
Specificity of the diagnosis of bacterial vs viral acute infection | 1 month
  Specificity of the diagnosis of bacterial vs viral acute infection using proposed method

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Y Hancharou, Dr, Study Director — Head of the Laboratory for Immunology and Cellular Biotechnology, The Republican Research and Practical Center for Epidemiology and Microbiology

IPD SHARING:
Plan to Share IPD: No